CLINICAL TRIAL: NCT06121713
Title: Effect of Green Coffee Extract Combined With Alpha-Lipoic Acid on Blood Glucose Homeostasis in Healthy Adults
Acronym: GCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Iovate Health Sciences International Inc (Industry)
Responsible Party: Principal Investigator, Jenna Gillen, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 44741
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GCE + Low ALA (Active Comparator): Green coffee extract and a low dose of alpha-lipoic acid prior to an oral glucose tolerance test
  Interventions: Dietary Supplement: GCE + Low ALA
- GCE + High ALA (Active Comparator): Green coffee extract and a moderate dose of alpha-lipoic acid prior to an oral glucose tolerance test
  Interventions: Dietary Supplement: GCE + High ALA
- Placebo (Placebo Comparator): Inert placebo pill prior to an oral glucose tolerance test
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GCE + Low ALA — Participants will consume a pill containing 200mg green coffee extract and 200mg alpha-lipoic acid 30 minutes before a 75g oral glucose tolerance test
  Arms: GCE + Low ALA
Dietary Supplement: GCE + High ALA — Participants will consume a pill containing 200mg green coffee extract and 400mg alpha-lipoic acid 30 minutes before a 75g oral glucose tolerance test
  Arms: GCE + High ALA
Dietary Supplement: Placebo — Participants will consume a placebo pill (500mg insoluble microcrystalline cellulose, 5mg magnesium stearate, 5mg silicon dioxide) prior to a 75g oral glucose tolerance test
  Arms: Placebo

SUMMARY:
Green coffee extract (GCE) supplementation has been shown to induce favourable health benefits on glucose metabolism and weight management. Previous literature suggests that the benefits of GCE are due to the high bioavailability of chlorogenic acid (CGA) which is known for its antioxidant and anti-inflammatory properties but is destroyed during the bean roasting process used to make coffee in Western societies. Whilst some studies examining chronic and high dose GCE supplementation (4-12 weeks) report beneficial effects on glucose metabolism and reductions in body mass following supplementation, comparably less is known about the effect of acute (single dose) GCE supplementation. Another natural compound, alpha-lipoic acid (ALA) has antioxidant properties and may also benefit glucose metabolism. The purpose of the current study is to determine the impact of acute supplementation of GCE with ALA on postprandial blood glucose concentration following consumption of a carbohydrate drink in healthy adults. A secondary objective is to evaluate the effect of GCE+ALA on blood insulin concentrations, insulin sensitivity, glucose oxidation, and perceptions of appetite.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine if GCE combined with ALA supplementation influences postprandial glucose metabolism. Participants will complete 3 visits to the investigator's laboratory at the University of Toronto. On each occasion, participants will consume a sugary drink (75g sugar) and investigators will take blood and breath samples for 2 hours. Participants will also be asked to fill out some questionnaires about appetite during this time. Thirty minutes before consuming the sugary drink, participants will consume one of the following pill supplements in a randomized order: 1) 200mg CGE + 200mg ALA; 2) 200mg GCE + 400mg ALA; or 3) Placebo (no CGE or ALA).

The study will advance knowledge regarding the effects of GCE and ALA on postprandial glycemia and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* BMI 20 - 30 kg/m2
* Weight stable (within ± 2kg for at least 6 months)
* Experiencing monthly menstrual periods (eumenorrheic) if female
* Non-smoker

Exclusion Criteria:

* Previous history of cardiovascular or metabolic disease
* Use of medication for managing blood glucose or lipid metabolism
* Current use of monophasic or biphasic oral contraceptives within the last 3 months (triphasic oral contraceptives are okay)
* Current supplementation of green coffee extract or supplementing in the last 3 months
* Irregular menstrual cycles (<21 days or >35 days)
* Pregnant or lactating
* Recreational smoking of any form (tobacco or cannabis)
* Not willing to consume the 24-hour control diet prior to metabolic trials

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Glucose incremental area under the curve | 2 hours
  glucose incremental area under the curve measured during an oral glucose tolerance test

SECONDARY OUTCOMES:
Mean glucose concentration | 2 hours
  Mean glucose concentration measured during an oral glucose tolerance test
Insulin incremental area under the curve | 2 hours
  insulin incremental area under the curve measured during an oral glucose tolerance test
Mean insulin concentration | 2 hours
  mean insulin concentration measured during an oral glucose tolerance test
peak glucose concentration | 2 hours
  peak glucose concentration measured during an oral glucose tolerance test
peak insulin concentration | 2 hours
  peak insulin concentration measured during an oral glucose tolerance test
Postprandial glucose oxidation | 2 hours
  Postprandial glucose oxidation measured with a metabolic tracer
Appetite perceptions | 2 hours
  Visual analog scales (0-100) will be used to determine perceptions of hunger, satisfaction, fullness, and prospective food consumption with higher scores denoting increased perceptions.
Insulin sensitivity | 2 hours
  insulin sensitivity measured via the Matsuda Index during an oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Gillen, PhD, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No